CLINICAL TRIAL: NCT01868776
Title: Effect of Buffered Lidocaine on the Success of the Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis
Brief Title: Effect of Buffered Numbing Solution on Patients With Toothaches
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Melissa Drum, Associate Professor, Ohio State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: buffered anesthetic toothache
Record Dates: First submitted 2013-05-30; First posted 2013-06-05 (Estimated); Results first posted 2015-05-29 (Estimated); Last update posted 2020-10-06 (Actual); Status verified 2020-09

CONDITIONS: Irreversible Pulpitis (Toothache)
MeSH Terms: conditions — Toothache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- buffered lidocaine (Experimental): 4% lidocaine with 1:100,000 epinephrine/0.18 mEq/mL sodium bicarbonate.
  Interventions: Drug: buffered lidocaine
- nonbuffered lidocaine (Active Comparator): 4% lidocaine with 1:100,000 epinephrine
  Interventions: Drug: nonbuffered lidocaine

INTERVENTIONS:
Drug: buffered lidocaine
  Arms: buffered lidocaine
Drug: nonbuffered lidocaine
  Arms: nonbuffered lidocaine

SUMMARY:
The purpose of this study is to determine the effect of buffered lidocaine (a numbing solution) on the ability to numb patients with toothaches. Buffered anesthetic (numbing) solutions have shown promise in some medical and dental research. Patients presenting with toothaches will be given either a buffered numbing solution or a nonbuffered numbing solution. Neither the patient nor the operator will know which solution they will receive. Root canal treatment will be performed on the tooth and the ability of the buffered versus non-buffered numbing solutions will be compared.

ELIGIBILITY:
Inclusion Criteria:

* patients with a diagnosis of irreversible pulpitis (toothache) in a mandibular posterior tooth (back/bottom tooth) with moderate to severe pain
* ages 18 -65 years of age
* in good health (ASA I or II)
* able to grant informed consent.

Exclusion Criteria:

* allergy to lidocaine (numbing solution
* significant medical problem (ASA III or IV)
* have taken CNS depressants or analgesic medications within the last 24 hours
* pregnancy or lactating
* non-English speaking
* inability to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Ohio State University College of Dentistry, Postle Hall, Columbus, Ohio, United States

REFERENCES:
- [Background] DiFazio CA, Carron H, Grosslight KR, Moscicki JC, Bolding WR, Johns RA. Comparison of pH-adjusted lidocaine solutions for epidural anesthesia. Anesth Analg. 1986 Jul;65(7):760-4. PMID 3717616
- [Background] Zahl K, Jordan A, McGroarty J, Sorensen B, Gotta AW. Peribulbar anesthesia. Effect of bicarbonate on mixtures of lidocaine, bupivacaine, and hyaluronidase with or without epinephrine. Ophthalmology. 1991 Feb;98(2):239-42. doi: 10.1016/s0161-6420(91)32311-x. PMID 2008283
- [Background] Sinnott CJ, Garfield JM, Thalhammer JG, Strichartz GR. Addition of sodium bicarbonate to lidocaine decreases the duration of peripheral nerve block in the rat. Anesthesiology. 2000 Oct;93(4):1045-52. doi: 10.1097/00000542-200010000-00028. PMID 11020760
- [Background] Richtsmeier AJ, Hatcher JW. Buffered lidocaine for skin infiltration prior to hemodialysis. J Pain Symptom Manage. 1995 Apr;10(3):198-203. doi: 10.1016/0885-3924(94)00124-4. PMID 7629414
- [Background] Burns CA, Ferris G, Feng C, Cooper JZ, Brown MD. Decreasing the pain of local anesthesia: a prospective, double-blind comparison of buffered, premixed 1% lidocaine with epinephrine versus 1% lidocaine freshly mixed with epinephrine. J Am Acad Dermatol. 2006 Jan;54(1):128-31. doi: 10.1016/j.jaad.2005.06.043. PMID 16384767
- [Background] Ackerman WE 3rd, Ware TR, Juneja M. The air-liquid interface and the pH and PCO2 of alkalinized local anaesthetic solutions. Can J Anaesth. 1992 Apr;39(4):387-9. doi: 10.1007/BF03009051. PMID 1314142

RESULTS

PARTICIPANT FLOW:
Groups:
- Buffered: buffered lidocaine
- Nonbuffered: nonbuffered lidocaine
Period: Overall Study
Arm/Group | Buffered | Nonbuffered
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Buffered | Nonbuffered | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (11.3) | 35.5 (10.7) | 35.1 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 18 | 21 | 39
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With Successful Anesthesia (% of Patients Able to Have Treatment Without Additional Anesthesia)
Time Frame: pain at time of treatment (after buffered versus nonbuffered numbing solution) average of 15 minutes after injection
Measure: Count of Participants; unit: Participants
Groups:
- Buffered Lidocaine: 4% lidocaine with 1:100,000 epinephrine/0.18 mEq/mL sodium bicarbonate.
  buffered lidocaine
- Nonbuffered Lidocaine: 4% lidocaine with 1:100,000 epinephrine
  nonbuffered lidocaine
Arm/Group | Buffered Lidocaine | Nonbuffered Lidocaine
Number analyzed (Participants) | 50 | 50
Participants | 16 | 20

2. Primary Outcome: Effect of Buffered Lidocaine on the Success of the Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis.
Description: 100 patients diagnosed with symptomatic irreversible pulpitis of a mandibular posterior tooth randomly received a conventional inferior alveolar nerve block (IAN) block using either 2.8 ml of 4% lidocaine with 1:100,000 epinephrine or 2.8 ml of 4% lidocaine with 1:100,000 epinephrine buffered with sodium bicarbonate in a double-blind manner. For the buffered solution, each cartridge was buffered with 8.4% sodium bicarbonate to produce a final concentration of 0.18 mEq/mL of sodium bicarbonate. Fifteen minutes after administration of the IAN block, profound lip numbness was confirmed and endodontic access was initiated. Success was determined as no or mild pain on access or instrumentation of the root canal. Higher numbers on the VAS are indicative of more pain and less success and the VAS scale ranged from 0 to 170 mm.
Time Frame: approximately 15 minutes after injection
Measure: Number; unit: percentage of participants
Arm/Group | Buffered Lidocaine | Nonbuffered Lidocaine
Number analyzed (Participants) | 50 | 50
percentage of participants | 32 | 40

ADVERSE EVENTS:
Arm/Group | Buffered | Nonbuffered
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 0/50 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No